CLINICAL TRIAL: NCT01489072
Title: Comparison of the Efficacy of Two Bolus Doses of Remifentanil on the Incidence of Coughing During Emergence of Anesthesia.
Brief Title: Efficacy of Two Bolus Doses of Remifentanil on the Incidence of Coughing During Emergence of Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NM 2012-002
Record Dates: First submitted 2011-12-05; First posted 2011-12-09 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Cough; Anesthesia
MeSH Terms: conditions — Cough | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil 0.25 mcg/kg (Experimental): Administration of a bolus dose of remifentanil 0.25 mcg/kg before emergence of a desflurane-based anesthesia
  Interventions: Drug: Remifentanil
- Remifentanil 0.5 mcg/kg (Active Comparator): Administration of a bolus dose of remifentanil 0.5 mcg/kg before emergence of a desflurane-based anesthesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Bolus dose of intravenous remifentanil 0.25 mcg/kg given once before emergence of general anesthesia
  Arms: Remifentanil 0.25 mcg/kg
Drug: Remifentanil — Bolus dose of intravenous remifentanil 0.5 mcg/kg given once before emergence of general anesthesia
  Arms: Remifentanil 0.5 mcg/kg

SUMMARY:
This study is designed to compare the effects of two bolus doses of intravenous remifentanil given prior to the emergence of anesthesia:

* on the incidence of perioperative coughing
* on the time needed for the emergence of a desflurane-based anesthesia
* on the incidence of sore throat after extubation.

The investigators hypothesis is that the use of a higher remifentanil bolus dose (0.5 mcg/kg) given prior to emergence of a desflurane-based anesthesia will reduce the incidence of perioperative coughing when compared to a lower dose of remifentanil (0.25 mcg/kg).

DETAILED DESCRIPTION:
Emergence is an important period of general anesthesia during which several problems can occur. Coughing, hypertension, tachycardia and agitation have been observed during emergence of general anesthesia.

Most patients will cough during emergence. Different techniques and drugs have been studied to reduce coughing during emergence.

There is some evidence supporting the administration of intravenous opioids prior to emergence of general anesthesia to reduce perioperative coughing, agitation and haemodynamic stimulation. However, depending on the type of opioids given, this may delay the emergence from anesthesia. The effect of a remifentanil infusion given in combination with isoflurane as the volatile agent has been shown to reduce the incidence of perioperative coughing without delaying the emergence of anesthesia. The effect of a small bolus of remifentanil given prior to emergence to prevent perioperative coughing has yet to be studied.

Desflurane is a newer volatile agent allowing early recovery from anesthesia. This agent has led to earlier discharge and more rapid resumption of normal activities after surgery. However, an incidence of coughing around 70% has been reported after a desflurane-based anesthesia.

This study will compare the effects of two bolus doses of remifentanil (0.25 mcg/kg to 0.5 mcg/kg) when given prior to emergence to prevent perioperative coughing after a desflurane-based anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Physical status 1-3
* Patients undergoing elective surgery under general anesthesia requiring endotracheal intubation (excluding head and neck surgery)

Exclusion Criteria:

* Current use of ACE inhibitors
* Chronic cough
* Asthma or severe pulmonary disease
* Pulmonary tract infection
* Anticipated difficult intubation
* Current use of opioids
* Current use of cough medicine
* Contraindication to remifentanil
* Pregnancy
* Symptomatic cardiac, renal or hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of coughing during emergence and the first ten minutes after extubation | From emergence until 10 minutes after extubation

SECONDARY OUTCOMES:
Time elapsed between the bolus dose of remifentanil and extubation | Assessed at emergence of general anesthesia
Incidence of sore throat one hour after extubation | Assessed one hour after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massicotte, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal-Hôpital Notre-Dame, Montreal, Quebec, Canada